CLINICAL TRIAL: NCT01282112
Title: Sedation for Brainstem Evoked Auditory Response (BEAR) Testing Using Intravenous Pentobarbital - A Retrospective Study
Brief Title: Sedation for Brainstem Evoked Auditory Response (BEAR) Testing Using Intravenous Pentobarbital
Status: Completed | Type: Observational
Sponsor: Akron Children's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 101014
Record Dates: First submitted 2011-01-21; First posted 2011-01-24 (Estimated); Last update posted 2014-06-26 (Estimated); Status verified 2014-06

CONDITIONS: Childrens 0 to 18 Years of Age Who Require Moderate Sedation

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a retrospective chart review study (700 charts from 2002 to 2010)of children from 0 to 18 years of age who have undergone Brainstem Evoked Auditory Response (BEAR)testing using midazolam and pentobarbital protocol for moderate sedation. The specific aims of this study are two-fold:

1. to determine the efficacy of intravenous pentobarbital during BEAR testing in the pediatric population using a standardized protocol; and
2. to evaluate the incidence of adverse events (major and minor), paradoxical reaction and failed sedation and identify predictors for failure and adverse events if any.

DETAILED DESCRIPTION:
Sedation Protocol:

* Versed: 0.1mg/kg IV
* Induction: 2mg/kg IV in children <1 year; 3mg/kg IV in children >1year
* Maintenance phase: 1mg/kg IV every 3 to 5 minutes with a maximal dose of 8mg/kg or 200 mg

Definition of terms:

* Failed Sedation: A case in which a patient is inadequately sedated after receiving maximum required dosages such that the test cannot be completed.
* Paradoxical Reaction: Also known as 'pentobarbital rage' is defined as a patient experiencing sustained, inconsolable, and severe irritability or combativeness. This can occur anywhere between 30 minutes after administration of pentobarbital to post recovery phase.
* Prolonged Sedation: A case in which either the patient cannot be discharged 3 hours after administration of the last sedating medication. It could also be a case in which patient is not back to baseline in 24 hours.
* Hypoxia: This is defined as a sustained decrease in oxygen saturation (>30 seconds) of more than 10% from baseline.
* Time to goal sedation: Time in minutes from initial administration of midazolam to the achievement of adequate sedation of the patient/start of procedure.
* Time to recovery: time in minutes from the last dose of pentobarbital to recovery of baseline status.
* Time to discharge: Time in minutes from administration of midazolam to discharge of patient from recovery room.

ELIGIBILITY:
Inclusion Criteria:

* Children from 0 to 18 years of age
* undergoing BEAR testing using midazolam and pentobarbital protocol for moderate sedation

Exclusion Criteria:

* Children greater that 18 years of age
* Patients with incomplete data

Max Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Children from 0 to 18 years of age undergoing BEAR testing using midazolam and pentobarbital protocol for moderate sedation.
Sampling Method: Non-Probability Sample
Enrollment: 416 (Actual)
Dates: Start 2011-01; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Determine the efficacy of intravenous pentobarbital during BEAR testing in the pediatric population using a standardized protocol. | 2002 through 2010
Evaluate the incidence of adverse events (major and minor) | 2002 through 2010

SECONDARY OUTCOMES:
Evaluate the incidence of paradoxical reaction | 2002 through 2010
Evaluate the incidence of failed sedation | 2002 through 2010
Identify predictors for failure and adverse events, if any | 2002 through 2010

CONTACTS AND LOCATIONS:
Overall Officials: Urmila Tirodker, MD, Principal Investigator — Akron Children's Hospital
Locations (1):
- Akron Children's Hospital, Akron, Ohio, United States

REFERENCES:
- [Background] Mason KP, Zurakowski D, Karian VE, Connor L, Fontaine PJ, Burrows PE. Sedatives used in pediatric imaging: comparison of IV pentobarbital with IV pentobarbital with midazolam added. AJR Am J Roentgenol. 2001 Aug;177(2):427-30. doi: 10.2214/ajr.177.2.1770427. PMID 11461876
- [Background] Mason KP, Zurakowski D, Connor L, Karian VE, Fontaine PJ, Sanborn PA, Burrows PE. Infant sedation for MR imaging and CT: oral versus intravenous pentobarbital. Radiology. 2004 Dec;233(3):723-8. doi: 10.1148/radiol.2333031872. Epub 2004 Oct 29. PMID 15516603
- [Background] Karian VE, Burrows PE, Zurakowski D, Connor L, Mason KP. Sedation for pediatric radiological procedures: analysis of potential causes of sedation failure and paradoxical reactions. Pediatr Radiol. 1999 Nov;29(11):869-73. doi: 10.1007/s002470050715. PMID 10552071
- [Background] Strain JD, Campbell JB, Harvey LA, Foley LC. IV Nembutal: safe sedation for children undergoing CT. AJR Am J Roentgenol. 1988 Nov;151(5):975-9. doi: 10.2214/ajr.151.5.975. PMID 3263031